CLINICAL TRIAL: NCT05707221
Title: Effect of Different Cleaning Regimes on Biofilm Formation of Acrylic Based Removable Orthodontic Appliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Dheaa Hussein Al-Groosh, Prof.Dr Dheaa Hussein Al-Groosh, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: cleaning of ROA
Record Dates: First submitted 2022-12-25; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Oral Disease
Keywords: Oral biofilm; Removable Orthodontic appliance; Cleaning Removable appliances
MeSH Terms: conditions — Mouth Diseases

STUDY DESIGN:
Intervention Model Description: The removable appliance will be assigned randomly and blindly and fitted into the oral cavity of the patient for one week. Each individual will be given a pack containing the cleansing pack and an instruction sheet describing the cleaning regimen for his/ her appliance. The packs are similar in shape and color and will be prepared by a third person who does not know the purpose of the study. The volunteer will be grouped into three groups:
  Group 1: patients will be instructed to brush both sides of the removable appliance once a day for 1 minute before bedtime using the denture brush and the CHX toothpaste (lacalut active, Germany) provided and water. Group 2: patients will be instructed to immerse the appliance in 150 ml cup with tap water and dissolve one cleansing (lacalut DENT cleaning tablet, Germany) tablet for 20 minutes according to the manufacture instructions. Group 3: Combination of brushing with CHX and cleaning tablets.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Sequence Generation: A computer random generator will be used to develop a simple randomization Allocation Concealment: This will be achieved using sequentially numbered, opaque and sealed envelopes which will be numbered according to the study numbers. Each envelope includes the treatment allocation card (group 1, 2 or 3) and the related cleaning method with instruction card.
  Blinding: An independent person will be responsible for giving the patient the envelope, all data collection and counting will be completed by a microbiologist who would not know about the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mechanical cleaning method by denture brush and Chlorhexidine toothpaste (Active Comparator): patients will be instructed to brush both sides of the removable appliance once a day for 1 minute before bedtime using the toothbrush and the CHX toothpaste provided and water
  Interventions: Other: cleaning removable acrylic appliance with denture brush and chlorhexidine toothpaste
- chemical cleaning method with cleaning tablet (Active Comparator): patients will be instructed to immerse the appliance in 150 ml cup with tap water and dissolve one cleansing tablet for 20 minutes according to the manufacture instructions.
  Interventions: Other: cleaning removable acrylic appliance with cleansing tablet
- combination of mechanical and chemical cleaning (Active Comparator): first submitted to the mechanical method, followed by the chemical method.
  Interventions: Other: combination of mechanical and chemical cleaning

INTERVENTIONS:
Other: cleaning removable acrylic appliance with denture brush and chlorhexidine toothpaste — mechanical cleaning of removable appliance by the patient for 7 days before bedtime for one minute
  Other Names: Denture brush (Foramen denture brush, Spain), CHX toothpaste(Lacalute Active, Germany)
  Arms: mechanical cleaning method by denture brush and Chlorhexidine toothpaste
Other: cleaning removable acrylic appliance with cleansing tablet — chemical cleaning by patient for 7 days with cleansing tablet
  Other Names: cleansing tablet (Lacalute cleansing tablet, Germany)
  Arms: chemical cleaning method with cleaning tablet
Other: combination of mechanical and chemical cleaning — cleaning the appliance with denture brush and CHX toothpaste followed by the cleansing tablet
  Other Names: cleaning with brushing then with the cleaning tablet
  Arms: combination of mechanical and chemical cleaning

SUMMARY:
This study is to evaluate the effects of different cleaning regimes i.e. chemical and mechanical on biofilm formation of an acrylic based removable orthodontic appliance and to find out if surface modification i.e. polished acrylic fitting surface, have an impact on cleaning the biofilm formation.

DETAILED DESCRIPTION:
It is double-blind, parallel, randomized clinical trial conducted in the orthodontic clinic after obtaining the ethical approval from the ethics committee of the department. Thirty nine orthodontic patients who meet the eligibility criteria will be included in the study and will be provided by the patient information sheet and consent form that will explain the nature of the study. After initial approval from the patient an alginate impression of the maxillary arch will be taken and a negative replica will be made by type IV stone. The wire framework of the removable appliance will be fabricated according to the design for the case. After applying a separating medium, an acrylic base will be fabricated using the orthodontic acrylic powder and liquid (Orthocryle, Dentaurum, Ispringen, German) with a ratio of (2.5 parts powder to 1 part liquid) according to the manufacturer's instruction with four wells on each side of the fitting surface of the appliance. Acrylic samples i.e. tiles of different surface texture will be made. An acrylic sheet of 1 mm thickness will be made using a mold material. One sheet will be polished using a conventional polishing technique until a glossy surface appears, whereas, the other sheet will be kept without modification. Tiles of 5mm in diameter will be bored using a trephine bur on both sides of the acrylic sheets and each set of tiles i.e. the polished and unpolished samples will be color coated from its seated surface. The acrylic tiles (5mm in diameter and 1mm thickness) will be placed and fixed into the holes created using sticky wax. The acrylic samples will be randomly seated, The appliance will be sterilized using proper sterilization protocol. The removable appliance will be assigned randomly and blindly and fitted into the oral cavity of the patient for one week. Each individual will be given by an independent person a pack containing the cleansing pack and an instruction sheet describing the cleaning regimen for his/ her appliance. The packs are similar in shape and color and will be prepared by a third person who does not know the purpose of the study. The participant will be grouped into three groups:

1. Brushing with denture brush and chlorhexidine (CHX) toothpaste (lacalut Active, Germany) for one minute.
2. Chemical cleaning i.e. Lacalut cleaning tablet (lacalut DENT cleaning tab, Germany), fill the cup to the marked line (150 mL) with tap water, dissolve one cleansing tablet and wait for 20 minutes then wash it with tap water.
3. Combination of brushing with CHX toothpaste and cleaning tablet. At the end of the study period, the acrylic samples will be removed carefully and applied into a petri dish containing PBS via a sterile tweezer. The samples will be then immersed twice in a 25ml sterile tubes containing PBS to remove the planktonic bacteria and inserted into 5ml bijou tube containing 1mm PBS. The sample will be vortex mixed for 1 minute to disseminate the biofilm and create a homogenous solution. Ten-fold serial dilutions will be carried out in PBS before the samples are plated onto blood agar (BA), to give the total anaerobic count, mitis salivarius agar (MS), a selective agar for streptococci spp. and Mannitol salt agar (MA) for Staphylococci spp. BA and MS plates will be incubated anaerobically for 2-4 days at 37ºC using anaerobic cabinet whereas the MA will be incubated for 2 days in aerobic condition. All organisms from both selective and nonselective agars will be distinguished by colony morphology and will be characterized by Gram reaction and other confirmatory tests: 1. Catalase testing 2. Coagulase testing

ELIGIBILITY:
Inclusion Criteria:

* Presence of full upper permanent dentition
* Well-aligned teeth or mild crowding (less than 3mm)
* No history of sensitivity to any ingredient contained in the cleaning materials
* Nonsmoker
* Caries free

Exclusion Criteria:

* Participant taking steroid-based or antibacterial mouthwash or broad-spectrum antibiotics
* Mouth breather
* Participant taking medication that reduces salivary flow
* Pregnant lactating female

Ages: 7 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Estimated)
Dates: Start 2022-04-17 (Actual); Primary Completion 2023-02-25 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
microbial evaluation between the three cleaning methods | 7 days
  numbers of streptococcus species, staphylococcus species and total anaerobic bacteria will be evaluated after isolation from acrylic discs and culture.

SECONDARY OUTCOMES:
microbial evaluation between the polished and unpolished acrylic discs | 7 days
  numbers of streptococcus species, staphylococcus species and total anaerobic bacteria will be evaluated after isolation from acrylic discs and culture.

CONTACTS AND LOCATIONS:
Overall Officials: Dheaa Al-Groosh, Ph.D, Study Director — University of Baghdad
Locations (1):
- Baghdad college of dentistry, Baghdad, Bab-Almuadham, Iraq

REFERENCES:
- [Background] Albanna RH, Farawanah HM, Aldrees AM. Microbial evaluation of the effectiveness of different methods for cleansing clear orthodontic retainers: A randomized clinical trial. Angle Orthod. 2017 May;87(3):460-465. doi: 10.2319/072916-585.1. Epub 2016 Nov 15. PMID 27845562
- [Background] Eichenauer J, Serbesis C, Ruf S. Cleaning removable orthodontic appliances: a survey. J Orofac Orthop. 2011 Oct;72(5):389-95. doi: 10.1007/s00056-011-0043-2. English, German. PMID 21990062
- [Background] Leao RS, Maior JRS, Lemos CAA, Vasconcelos BCDE, Montes MAJR, Pellizzer EP, Moraes SLD. Complications with PMMA compared with other materials used in cranioplasty: a systematic review and meta-analysis. Braz Oral Res. 2018 Jun 7;32:e31. doi: 10.1590/1807-3107bor-2018.vol32.0031. PMID 29898018
- [Background] Lima EM, Moura JS, Del Bel Cury AA, Garcia RC, Cury JA. Effect of enzymatic and NaOCl treatments on acrylic roughness and on biofilm accumulation. J Oral Rehabil. 2006 May;33(5):356-62. doi: 10.1111/j.1365-2842.2005.01564.x. PMID 16629894
- [Background] Pathak AK, Sharma DS. Biofilm associated microorganisms on removable oral orthodontic appliances in children in the mixed dentition. J Clin Pediatr Dent. 2013 Spring;37(3):335-9. doi: 10.17796/jcpd.37.3.92230h6256v8697t. PMID 23855182
- [Background] Puri G, Berzins DW, Dhuru VB, Raj PA, Rambhia SK, Dhir G, Dentino AR. Effect of phosphate group addition on the properties of denture base resins. J Prosthet Dent. 2008 Oct;100(4):302-8. doi: 10.1016/S0022-3913(08)60210-3. PMID 18922259
- [Background] Rodriguez-Renteria M, Marquez-Preciado R, Ortiz-Magdaleno M, Bermeo-Escalona J, Sanchez-Vargas LO. Frequency of Pathogenic Microorganisms in Removable Orthodontic Appliances and Oral Mucosa in Children. J Clin Pediatr Dent. 2021 Apr 1;45(2):135-139. doi: 10.17796/1053-4625-45.2.11. PMID 33951170
- [Background] Schwindling FS, Rammelsberg P, Stober T. Effect of chemical disinfection on the surface roughness of hard denture base materials: a systematic literature review. Int J Prosthodont. 2014 May-Jun;27(3):215-25. doi: 10.11607/ijp.3759. PMID 24905261
- [Background] Xiao J, Moon Y, Li L, Rustchenko E, Wakabayashi H, Zhao X, Feng C, Gill SR, McLaren S, Malmstrom H, Ren Y, Quivey R, Koo H, Kopycka-Kedzierawski DT. Candida albicans Carriage in Children with Severe Early Childhood Caries (S-ECC) and Maternal Relatedness. PLoS One. 2016 Oct 14;11(10):e0164242. doi: 10.1371/journal.pone.0164242. eCollection 2016. PMID 27741258
- [Derived] Khawwam SI, Al-Groosh DH. Effect of Different Cleaning Regimes on Biofilm Formation of Acrylic-Based Removable Orthodontic Appliance: A Randomized Clinical Trial. ScientificWorldJournal. 2023 Oct 12;2023:9920850. doi: 10.1155/2023/9920850. eCollection 2023. PMID 37868294

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-12-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT05707221/Prot_SAP_ICF_000.pdf